CLINICAL TRIAL: NCT04761497
Title: Effects of Group Music Therapy Interventions on Alzheimer's Disease Patients: a Three-arm Randomized Controlled Blind Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, María Gómez-Gallego, Profª Dr María Gómez-Gallego, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PIC06/19
Record Dates: First submitted 2021-02-12; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; cognition.; behaviour; function; motor function; active music therapy; passive music therapy
MeSH Terms: conditions — Alzheimer Disease; Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- active music therapy (Experimental): Each session consisted of: song of welcome (patients had to greet and introduce themselves), rhythmic exercise (three songs were used; therapist and patients kept rhythm by clapping their hands), dance exercises (three songs were used; patients should make free body movements in response to music), game of recognition of songs and interpreters (four songs were used) and song of goodbye.
  Interventions: Other: Actice music therapy
- passive music therapy (Experimental): The therapist and the patients were seat listening to the music recorded in a CD. The therapist told patients which the name and the interpreter of each song of the list.
  Interventions: Other: Passive music therapy
- control (Placebo Comparator): Patients were watching nature videos for the same duration than the interventions. A therapist was with them facilitating the activity.
  Interventions: Other: Watching nature videos

INTERVENTIONS:
Other: Actice music therapy — active music therapy sessions for three months
  Arms: active music therapy
Other: Watching nature videos — nature videos sessions for three months
  Arms: control
Other: Passive music therapy — passive music therapy for three months
  Arms: passive music therapy

SUMMARY:
The purpose of this study is to determine what type of music therapy (active versus passive) approach has higher effects on clinical symptoms in advanced Alzheimer's disease patients

DETAILED DESCRIPTION:
Ninety AD patients from six nursing homes participated in the study. Nursing homes were randomly and blindly assigned to receive for three months either active music intervention, passive music listening or usual care. Effects on cognition, behaviour, daily living activities and motor function were assessed after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Nursing-home dwelling
* Diagnosis of probable Alzheimer's disease
* Mild or moderate stage (Clinical Classification of the Dementia)

Exclusion Criteria:

* Aphasia
* Hearing impairment that may affect participation in the activities.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2019-01-07 (Actual)

PRIMARY OUTCOMES:
Mini Examination of the Mental State | 0-3 months
  Cognitive status. Range 0-30. Higher scores indicate better cognition
Neuropsychiatric Inventory | 0-3 months
  Behavioural disorders. Range 0-144. Higher scores indicate greater behavioural problems
Geriatric depression scale | 0-3 months
  Mood status. Range 0-15. Higher scores indicate worse mood status
Barthel index | 0-3 months
  Functional status. Range 0-100.Higher scores indicate worse functional status
Tinneti scale.Higher scores indicate better motor function | 0-3 months. Range 0-28
  Motor function

CONTACTS AND LOCATIONS:
Locations (1):
- UCMurcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No